CLINICAL TRIAL: NCT02481323
Title: Preventing Cognitive Decline and Dementia From Cerebral Small Vessel Disease
Brief Title: Lacunar Intervention Trial 1 (LACI-1)
Acronym: Prevent-SVD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: PrevSVD-2015; 2015-001953-33 (EudraCT Number); 252 (AS-PG-14-033) (Other Grant/Funding Number: Alzheimer's Society UK)
Record Dates: First submitted 2015-06-19; First posted 2015-06-25 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Small Vessel Diseases; Cognitive Impairment; Stroke
Keywords: cerebral small vessel disease; cerebrovascular reactivity; cilostazol; isosorbide mononitrate
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction; Stroke | interventions — isosorbide-5-mononitrate; Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Active Comparator): Isosorbide mononitrate 25mg bd
  Interventions: Drug: isosorbide mononitrate
- Group 2 (Active Comparator): Cilostazol 100mg bd
  Interventions: Drug: cilostazol
- Group 3 (Active Comparator): Isosorbide mononitrate 25mg bd and cilostazol 100mg bd start immediately
  Interventions: Drug: isosorbide mononitrate; Drug: cilostazol
- Group 4 (Other): Isosorbide mononitrate 25mg bd and cilostazol 100mg bd delayed start
  Interventions: Drug: isosorbide mononitrate; Drug: cilostazol

INTERVENTIONS:
Drug: isosorbide mononitrate — slow release nitric oxide donor that enhances vasodilation and widely used in angina prophyaxis
  Other Names: Isotard
  Arms: Group 1; Group 3; Group 4
Drug: cilostazol — phosphodiesterase 3-inhibitor that enhances vessel wall function with weak antiplatelet effects
  Other Names: pletal
  Arms: Group 2; Group 3; Group 4

SUMMARY:
Phase II pilot randomised, factorial, short term dose escalation, open label, blinded intermediary endpoint trial, in two hospital centres in the UK, of tolerability and safety of cilostazol, isosorbide mononitrate, both or neither in patients with small vessel disease manifest as symptomatic small subcortical stroke.

DETAILED DESCRIPTION:
A quarter of all ischaemic strokes are lacunar (small vessel) in type, about 35000 per annum in the United Kingdom, and due to an intrinsic, non-atheromatous, non-cardioembolic perforating cerebral arteriolar disease. 'Small vessel disease' also affects the brain diffusely, causing up to 40% of dementias, alone or mixed with Alzheimer's disease, 350,000+ patients estimated currently in the United Kingdom. There is no proven treatment: conventional antiplatelet drugs may be ineffective or even hazardous, antihypertensive treatment and statins have been disappointing. The disease mechanism is poorly understood but endothelial dysfunction, blood-brain barrier failure and vessel stiffness appear to contribute to the pathogenesis. Promising data available for licensed drugs with relevant modes of action, cilostazol (>6000 stroke patients in the Asia Pacific region) and isosorbide mononitrate (ISMN, widely used in cardiac disease) support their testing in small vessel disease. This trial will be a phase 2, randomised, dose-escalation, factorial trial to test short-term administration of cilostazol, Isosorbide Mononitrate, both, or neither, to provide data on patient tolerability of dose (including headache, dizziness), safety (including blood pressure, platelet function), provide mechanistic evidence of efficacy (cerebrovascular reactivity, arterial compliance), and to inform the design of a larger phase 2-3 trial. The trial will recruit 60 patients with small vessel disease, in two expert stroke centres (Edinburgh and Nottingham) where there are suitable patients, expert stroke centres, established trials infrastructures and neuroimaging and platelet testing expertise. The trial will also advance methods to stratify patients by small vessel disease burden in routine practise and data on intermediary mechanistic outcomes to assist in planning future trials testing novel agents for either stroke or dementia.

ELIGIBILITY:
Inclusion Criteria:

* Mild symptomatic ischaemic stroke in the past four years compatible with a clinical lacunar stroke syndrome, with brain magnetic resonance imaging or computed tomography scanning that is compatible with a symptomatic small subcortical (lacunar) infarct, or if no recent relevant infarct is visible, that excluded other cause for symptoms
* Age > 35 years
* Independent in activities of daily living (modified Rankin ≤2)
* Able to give consent themselves

Exclusion Criteria:

* Other significant active neurological illness present since suffering stroke (eg seizures, multiple sclerosis, brain tumour)
* Age < 35
* Montreal Cognitive Assessment score <26
* Requiring assistance with activities of daily living (Modified Rankin ≥3)
* Active cardiac disease (atrial fibrillation, myocardial infarction in past 6 months, active angina, symptomatic cardiac failure)
* Carotid stenosis > 50% in the symptomatic artery territory requiring carotid endarterectomy (prior and apparently successful carotid endarterectomy is not an exclusion criterion)
* Definite indication for, or definite contraindication to either trial drug
* Unable to swallow
* Bleeding tendency (platelets<100, taking anticoagulant medication)
* Unlikely to comply with trial medication
* Planned surgery during the trial period
* History of intracranial haemorrhage (subdural haematoma, subarachnoid haemorrhage, intracerebral haemorrhage, but not asymptomatic haemorrhagic transformation of infarction)
* Other life threatening illness
* History of drug overdose or attempted suicide or significant active mental illness
* Pregnancy
* If recruited in Edinburgh and participating in cerebrovascular reactivity arm of trial: active respiratory illness (such as moderate to severe asthma or chronic obstructive airways disease), unable to tolerate magnetic resonance imaging or unable to lie flat

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Tolerability proportion of patients able to tolerate the target dose | 8 weeks
  proportion of patients able to tolerate the target dose

SECONDARY OUTCOMES:
Safety - bleeding | 12 weeks
  systemic or intracranial bleeding
Safety - recurrent stroke | 12 weeks
  recurrent vascular events,
Safety - death | 12 weeks
  death
Safety - blood pressure | 8 weeks
  reduction in blood pressure
Safety - bleeding | 8 weeks
  effect on platelet function assessed using p-selectin
Efficacy - cerebrovascular function | 8 weeks
  effect on cerebrovascular reactivity assessed using carbon dioxide challenge in magnetic resonance imaging
Efficacy - systemic arterial stiffness | 8 weeks
  effect on systemic large artery stiffness assessed with pulse wave velocity measurement
Tolerability Proportion of patients with headache that interferes with daily activities | 8 weeks
  Proportion of patients with headache that interferes with daily activities
Tolerability Proportion of patients with dizziness that interferes with daily activities | 8 weeks
  Proportion of patients with dizziness that interferes with daily activities
Tolerability Proportion of patients with nausea that interferes with daily activities | 8 weeks
  Proportion of patients with nausea that interferes with daily activities
Tolerability Proportion of patients with palpitations | 8 weeks
  Proportion of patients with palpitations
Tolerability Proportion of patients with loose stools | 8 weeks
  Proportion of patients with loose stools
Tolerability Tablet count | 8 weeks
  Tablet count

CONTACTS AND LOCATIONS:
Overall Officials: Joanna M Wardlaw, MD, Principal Investigator — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - University of Edinburgh, Edinburgh
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blair GW, Janssen E, Stringer MS, Thrippleton MJ, Chappell F, Shi Y, Hamilton I, Flaherty K, Appleton JP, Doubal FN, Bath PM, Wardlaw JM. Effects of Cilostazol and Isosorbide Mononitrate on Cerebral Hemodynamics in the LACI-1 Randomized Controlled Trial. Stroke. 2022 Jan;53(1):29-33. doi: 10.1161/STROKEAHA.121.034866. Epub 2021 Dec 1. PMID 34847709